# **OFFICIAL TITLE OF STUDY:**

Statewide Implementation of CAPABLE-Community Aging in Place, Advancing Better Living for Elders in the Michigan Medicaid Home and Community Based Waiver Program

> NCT NUMBER: NCT03634033 Registered August 16, 2018

**DOCUMENT DATE: JANUARY 29, 2020** 



## **Research Study**

**Title:** Statewide Implementation of CAPABLE (Community Aging-in-Place, Advancing Better Living for Elders) in the Michigan Medicaid Home and Community Based Waiver Program (NIA1R15AG058193-01A1S1; NCT03634033 Registered August 16, 2018)

You are being asked to participate in a research study. The box below highlights key information about this study for you to consider when making your decision whether or not to participate. Carefully consider the information on this form. Please ask questions about any information you do not understand before you decide whether to participate.

## **Key Information for You to Consider**

**Voluntary Consent.** You are being asked to volunteer for this research study. It is up to you whether you choose to participate or not. If you choose NOT to participate, do not sign this form.

**Purpose**. This is a collaborative research effort between the Grand Valley State University, the State of Michigan Department of Health and Human Services, and the National Institutes of Aging to find out if a toolkit for caregivers will help provide CAPABLE to participants.

**Duration**. It is expected that your participation will last one month.

**Procedures and Activities.** You will complete online surveys and training on use of the toolkit for caregivers. **Risks**. It is not expected that you will be placed at any physical, financial, or legal risk or harm to your employment status as a result of taking part in this study.

**Benefits**. There are no direct benefits to you, but we believe the knowledge gained from this study will increase clinician knowledge regarding CAPABLE and assist caregivers to care for their participants. **Alternatives**. If you choose to NOT participate, your employment will not be affected.

## How will this study help me?

Information from this study may help researchers understand how to help caregivers use a toolkit to assist participants to use CAPABLE and increase clinician knowledge regarding the toolkit. You will conduct CAPABLE with your participants with Alzheimer's Disease and Dementia and provide the toolkit to caregivers; in addition to "usual" waiver care services.

## Who can participate?

We are inviting all clinicians employed at waiver sites in Michigan.

## What will you receive?

If you agree to take part of the study you will complete online:

- Survey (5 minutes) asking you about your characteristics and work in the waiver.
- Training (1-hour) on use of the toolkit with caregivers.
- Survey about knowledge uptake (10-minutes).

#### What information will be used for research?

We will be collecting your data in an online survey platform (Qualtrics) on your characteristics and waiver work. We will have your name to follow your progress, but your name is known ONLY to the researcher and will be stored on a secure server. To prevent your identity to be connected with your data, we will remove your

name from the data. NO private information will be shared with anyone other than the researcher, and your results will be pooled among the other participants.

#### Are there risks?

It is not expected that you will be placed at any physical, financial, or legal risk or harm to your employment status as a result of taking part in this study. A Certificate of Confidentiality has been obtained from the Department of Health and Human Services for this study. To help protect your privacy, this certificate prevents researchers from being required (subpoenaed) to disclose identifying sensitive information collected for this study for use in court in most cases.

## What if I change my mind during the study?

You are free to not answer any survey question that makes you uncomfortable. You are also free to change your mind at any time and you may withdraw from the study if you like by calling Sandra Spoelstra at 616-331-5905. We will remove your data from our study.

# Who to call if you have questions?

If you have questions about the study, call: Sandra Spoelstra, Grand Valley State University, at 616-331-5905.

If you have any questions about your rights as a research participant, please contact the Office of Research Compliance & Integrity at Grand Valley State University, 1 Campus Dr., Allendale, MI Phone 616-331-3197. E-mail: rci@gvsu.edu

## What do I have to do?

If you are willing to participate, please type your name in the box below and complete the online surveys and training.

If you choose to not participate, exit out of this form.

This study was approved by the Grand Valley State University Human Research Review Committee (Protocol 20-213-H) on 2/19/2020.